CLINICAL TRIAL: NCT07142707
Title: A Randomized, Double-blind, Placebo-controlled First-in-human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Doses of MBX 4291 in Adult Participants With Obesity
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MBX 4291 in Adult Participants With Obesity
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MBX Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MBX-4O3001
Record Dates: First submitted 2025-08-04; First posted 2025-08-27 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-09

CONDITIONS: Obesity
Keywords: Body Weight; Body Mass Index; Overweight; Nutrition Disorders
MeSH Terms: conditions — Obesity; Body Weight; Overweight; Nutrition Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MBX 4291 (Part A) (Experimental): Participants will be administered single ascending doses of MBX 4291, or matching placebo.
  Interventions: Drug: MBX 4291
- MBX 4291 (Part B) (Experimental): Participants will be administered multiple ascending doses of MBX 4291, or matching placebo.
  Interventions: Drug: MBX 4291
- Placebo (Placebo Comparator): Participants will be administered single or multiple ascending doses of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MBX 4291 — MBX 4291 will be administered subcutaneously (SC)
  Arms: MBX 4291 (Part A); MBX 4291 (Part B)
Drug: Placebo — Placebo: Placebo will be administered subcutaneously (SC)
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single and multiple subcutaneous (SC) doses of MBX 4291 in adults with obesity.

DETAILED DESCRIPTION:
This is a Phase 1, double-blind, placebo-controlled first-in-human study to evaluate the single ascending doses (SAD) and multiple ascending doses (MAD) of MBX 4291 in participants with obesity, who are otherwise generally healthy. Approximately 64 patients aged 18 to 65 years old will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age of >18 to ≤65 years at the time of signing the informed consent.
* Has a BMI of ≥30 to <40 kg/m2 at screening and baseline.
* Weight-stable, i.e., no more than ±5% change in body weight for at least 3 months prior to screening and between screening and baseline.

Exclusion Criteria:

* History of, or currently active, significant illness or medical disorders that in the opinion of the investigator may preclude participants from participating in the study.
* History of currently active pancreatitis, type I and type II diabetes.
* Secondary causes of obesity, including but not limited to hypothalamic, monogenic, syndromic, or endocrine causes.
* A personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events (TEAEs) | The total duration of study participation for each participant including screening, treatment period, follow-up, and end of study visit will be up to 91 days in Part A and up to 99 days in Part B.

CONTACTS AND LOCATIONS:
Locations (1):
- MBX Biosciences Investigational Site, Knoxville, Tennessee, United States